CLINICAL TRIAL: NCT03933735
Title: A Multicenter, Phase 1, Open-label, Dose-escalation and Expansion Study of TNB-383B, a Bispecific Antibody Targeting BCMA in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of TNB-383B in Participants With Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNB383B.0001; 2023-506993-11 (Other: EU CT)
Record Dates: First submitted 2019-04-26; First posted 2019-05-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; TNB-383B
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm A: Dose Escalation (Experimental): Up to 15 cohorts of participants receiving sequentially ascending doses of TNB-383B are planned until maximum tolerated dose is reached or recommended phase 2 dose is identified.
  Interventions: Drug: TNB-383B
- Arm B: Dose Expansion Dose A (Experimental): An expansion cohort will be enrolled at the recommended phase 2 Dose A.
  Interventions: Drug: TNB-383B
- Arm B: Dose Expansion Dose B (Experimental): An expansion cohort will be enrolled at the recommended phase 2 Dose B.
  Interventions: Drug: TNB-383B
- Arm E: Monotherapy Once Every 4 Weeks (Q4W) (Experimental): An expansion cohort will be enrolled at the recommended phase 2 Dose A.
  Interventions: Drug: TNB-383B
- Arm F: Monotherapy Dose C (Experimental): An expansion cohort will be enrolled at the recommended phase 2 Dose C.
  Interventions: Drug: TNB-383B

INTERVENTIONS:
Drug: TNB-383B — Intravenous (IV) Injection

SUMMARY:
This is a phase 1, open-label study evaluating the safety, clinical pharmacology and clinical activity of TNB-383B, a BCMA x CD3 T-cell engaging bispecific antibody, in participants with relapsed or refractory MM who have received at least 3 prior lines of therapy. The study consists of 4 portions, a monotherapy dose escalation (Arm A) and a monotherapy dose expansion (Arm B), Monotherapy once every 4 weeks (Q4W) dosing (Arm E), Monotherapy once every 3 weeks (Q3W) dosing (Arm F). Arm A will evaluate the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) profiles of escalating doses of single-agent TNB-383B, administered Q3W, in approximately 73 participants. Once the maximum tolerated dose (MTD) or recommended phase 2 dose, (RP2D) is identified in Arm A, Arm B will be initiated to further characterize the safety, tolerability, PK and PD profiles of the MTD/RP2D 2 dose expansion arms of 48 participants each. Dose A will be evaluated as a monotherapy Q4W, in Arm E to further characterize the safety, tolerability, PK and PD profiles of the MTD/RP2D 2 dose expansion arms of 20 participants. Dose C will be evaluated as a monotherapy, in Arm F to further characterize the safety, tolerability, PK and PD profiles of the MTD/RP2D 2 dose expansion arms of 25 participants.

ELIGIBILITY:
Inclusion Criteria:

* Has received three or more prior lines of therapy with exposure to a proteasome inhibitor (PI), an immunomodulatory imide (IMiD) and an anti-CD38 monoclonal antibody.
* Must have adequate bone marrow function as defined in the protocol.
* Must have an estimated glomerular filtration rate >= 30 mL/min as estimated by the Modification of Diet in Renal Disease formula.
* Must have total bilirubin <= 1.5 × upper limit of normal ([ULN]; except if the subject has a known diagnosis of Gilbert's syndrome, in which case bilirubin must be < 3 x ULN).
* Serum calcium (corrected for albumin) at or below the ULN range.
* Has Measurable Disease, defined as at least 1 of the following:

  * Serum M-protein >= 0.5 g/dL (>= 5 g/L).
  * Urine M-protein >= 200 mg / 24h.
  * Serum free light chain (FLC) assay: Involved FLC level >= 10 mg/dl (>=100 mg/L) and an abnormal serum FLC ratio (< 0.26 or > 1.65).
* Has confirmed evidence of relapse/progression from the immediately prior MM therapy, or participant is relapsed/refractory to the immediately prior MM therapy.
* Consents to a fresh pretreatment bone marrow tumor biopsy or has adequate archival bone marrow tumor tissue that was collected within 6 months prior to screening and without intervening treatment.

Exclusion Criteria:

* Has been diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of basal cell or squamous cell carcinoma of the skin, in situ malignancy, low-risk prostate carcinoma after curative therapy, or complete resection/curative therapy of an advanced malignancy.
* History of central nervous system involvement by their myeloma.
* History of Grade >= 3 peripheral neuropathy.
* History of plasma cell leukemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes (POEMS) syndrome, or amyloidosis.
* Has received another investigational drug within 21 days of enrollment.
* Has ever received BCMA-targeted therapy.
* Has received a autologous stem cell transplant within 12 weeks or an allogeneic stem cell transplant within 1 year of the first dose of study drug treatment.
* Has any medical or psychiatric condition which in the opinion of the investigator or study Medical Monitor places the participant at an unacceptably high risk for toxicities, could interfere with successful or safe delivery of therapy, or could interfere with evaluation of the investigational product or interpretation of participant safety or study results.
* Has received any therapy to treat cancer or undergone a major surgical procedure within 21 days, or within 5 half-lives of an anticancer drug, prior to the first dose of study treatment, whichever is shorter.
* Has known active infection Grade >= 2 requiring anti-infective treatment.
* Has a history of major cardiac abnormalities.
* Has unresolved adverse events as defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting toxicities (DLT) | Day 21
  A DLT is defined as a Treatment-emergent adverse event that is not unequivocally due to the participant's underlying malignancy or other extraneous cause.
Number of Participants with Adverse Events (AEs) and/or Serious Adverse Events (SAEs) | Up to 3 Years
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Maximum Observed Plasma Concentration of TNB-383B (Cmax) | Week 12
  Cmax of TNB-383B.
Time to Cmax of TNB-383B (Tmax) | Week 12
  Time to maximum plasma concentration (Tmax) of TNB-383B.
Area Under the Concentration Versus Time Curve from Time Zero to the Last Measurable Concentration (AUClast) | Week 12
  Area under the concentration versus time curve from time zero to the last measurable concentration of TNB-383B.
Clearance (CL) of TNB-383B | Week 12
  Clearance is defined the volume of plasma cleared of the drug per unit time.
Terminal Phase Elimination Rate Constant (Beta) of TNB-383B | Week 12
  Apparent terminal phase elimination rate constant of TNB-383B.
Terminal Half-Life (t1/2) of TNB-383B | Week 12
  Terminal half-life (t1/2) of TNB-383B.
Number of Participants with of Anti-drug Antibody (ADA) | Up to Month 48
  The number of participants with anti-TNB-383B antibodies.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to Month 48
  ORR is defined as confirmed Stringent complete response (sCR) + Complete response (CR) + very good partial response + partial response [PR]).
Percentage of Participants with Overall Survival (OS) | Up to 48 Months
  OS is defined as time from the first dose of TNB-383B to the date of death, from any cause.
Percentage of Participants with Progression-Free Survival (PFS) | Up to 48 Months
  Progression-free survival time is defined as the time from the first dose of TNB-383B to progression or death, whichever occurs first.
Time-to-Progression (TTP) | Up to 48 Months
  TTP is defined as the time from the first dose of TNB-383B to the date of the first documented disease progression.
Time-to-Response (TTR) | Up to 48 Months
  TTR is defined as the time from the first dose of TNB-383B to the date of the first assessment having documented the response.
Duration of Objective Response (DOR) | Up to 48 Months
  DOR is defined as the time from the initial objective response to disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (14):
- United States (10):
  - University of California San Francisco (UCSF) - Parnassus Heights /ID# 238680, San Francisco, California
  - Tulane University School of Medicine /ID# 242322, New Orleans, Louisiana
  - Mayo Clinic - Rochester /ID# 238683, Rochester, Minnesota
  - Washington University-School of Medicine /ID# 238681, St Louis, Missouri
  - Mt Sinai /ID# 242317, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 244831, New York, New York
  - University of North Carolina /ID# 238685, Chapel Hill, North Carolina
  - Atrium Health Levine Cancer Institute /ID# 238786, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 238787, Winston-Salem, North Carolina
  - Wisconsin Medical Center /ID# 238684, Milwaukee, Wisconsin
- Germany (4):
  - Universitaetsklinikum Koeln /ID# 239676, Cologne, North Rhine-Westphalia
  - Duplicate_Universitaetsklinikum Muenster /ID# 239637, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 239638, Dresden, Saxony
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 239636, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Souza A, Shah N, Rodriguez C, Voorhees PM, Weisel K, Bueno OF, Pothacamury RK, Freise KJ, Yue S, Ross JA, Polepally AR, Talati C, Lee S, Jin Z, Buelow B, Vij R, Kumar S. A Phase I First-in-Human Study of ABBV-383, a B-Cell Maturation Antigen x CD3 Bispecific T-Cell Redirecting Antibody, in Patients With Relapsed/Refractory Multiple Myeloma. J Clin Oncol. 2022 Nov 1;40(31):3576-3586. doi: 10.1200/JCO.22.01504. Epub 2022 Aug 27. PMID 36029527